CLINICAL TRIAL: NCT07211061
Title: A SIX WEEK CLINICAL STUDY TO EVALUATE THE EFFECT OF A REGIMEN ON GINGIVITIS
Brief Title: A Study is to Evaluate a Regimen on Gingivitis Using Traditional and Novel Assessment Methods
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011068
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Cetylpyridinium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Hygiene Regimen (Experimental): toothpaste, electric toothbrush, and mouth rinse
  Interventions: Drug: Stannous Fluoride Dentifrice; Device: electric toothbrush; Drug: Cetylpyridinium Chloride (CPC)
- Negative Control (Active Comparator): toothpaste and manual toothbrush
  Interventions: Drug: Sodium Fluoride Dentifrice; Device: manual toothbrush

INTERVENTIONS:
Drug: Stannous Fluoride Dentifrice — brush 2x a day in using a power brush (2 minutes of brushing)
  Arms: Oral Hygiene Regimen
Drug: Sodium Fluoride Dentifrice — brush in their customary manner
  Arms: Negative Control
Device: electric toothbrush — brush using a electric brush (2 minutes of brushing)
  Arms: Oral Hygiene Regimen
Drug: Cetylpyridinium Chloride (CPC) — use 20 ml of mouth rinse for 30 seconds
  Arms: Oral Hygiene Regimen
Device: manual toothbrush — brush in their customary manner
  Arms: Negative Control

SUMMARY:
Subjects who have shown evidence of gingivitis and plaque will be enrolled in this study. Each subject will be randomly assigned to one of two treatment products. The regimen group will be asked to brush 2x a day in using a power brush (2 minutes of brushing), followed by using 20 ml of mouth rinse for 30 seconds for 6 weeks. The negative control group will be asked to brush 2x a day using a manual toothbrush in their customary manner for 6 weeks. Oral Soft Tissue (OST) assessments, gingivitis and plaque measurements will be taken at 4 time-points: Baseline (BL); Week 1; Week 3; and Week 6.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent to participate in the study;
* Be 18 years of age or older;
* Agree not to participate in any other oral/dental product studies during the course of this study;
* Agree to delay any elective dentistry (including dental prophylaxis) until the study has been completed;
* Agree to refrain from any form of non-specified oral hygiene during the treatment periods, including but not limited to the use of products such as floss or whitening products;
* Have a Baseline MGI score of at least 1.75 but not greater than 2.3;
* Have at least 20 bleeding sites (sites with a score of 1 or 2 on the GBI index);
* Agree to return for all scheduled visits and follow study procedures;
* Be in good general health, as determined by the Investigator/designee based on a review of the health history/update for participation in the study.

Exclusion Criteria:

* Have had a dental prophylaxis within 2 weeks of Baseline visit;
* Have taken antibiotics or used anti-gingivitis / anti-bacterial oral care products such as chlorhexidine or Listerine within 2 weeks of plaque sampling visits;
* Have rampant caries, open or untreated caries, severe gingivitis, or advanced periodontitis requiring prompt treatment; or,
* Need an antibiotic prophylaxis prior to dental visits,
* Present with any disease or condition(s) that could be expected to interfere with examination procedures or the subject's safe completion of the study,
* Are pregnant (Self-reported) or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-09-21 (Actual); Primary Completion 2011-11-10 (Actual); Study Completion 2011-11-10 (Actual)

PRIMARY OUTCOMES:
Bleeding (GBI) | Week 1, Week 3, and Week 6
  Gingival Bleeding Index- evaluation of bleeding from gingival tissue, score from 0-2

SECONDARY OUTCOMES:
Inflammation (MGI) | Week 1, Week 3, and Week 6
  Modified Gingival Index- evaluation of the level of gingival tissue inflammation, scores from 0-4

CONTACTS AND LOCATIONS:
Locations (1):
- Bio-Sci Research (Out of Business), Las Vegas, Nevada, United States